CLINICAL TRIAL: NCT06304571
Title: A Phase I, Open-label, Dose-Escalation and Dose-expansion Clinical Trial to Evaluate the Safety, Tolerability, Pharmacokinetics, Immunogenicity and Efficacy of HC006 in Advanced Solid Tumor Subjects
Brief Title: A Study of HC006 in Subjects With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: HC Biopharma Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HC006-001
Record Dates: First submitted 2024-03-05; First posted 2024-03-12 (Actual); Last update posted 2025-05-06 (Actual); Status verified 2025-04

CONDITIONS: Advanced Solid Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- HC006 Dose Escalation (Experimental)
  Interventions: Drug: HC006
- HC006 Dose Expansion (Experimental)
  Interventions: Drug: HC006

INTERVENTIONS:
Drug: HC006 — Specified dose on specified days

SUMMARY:
The purpose of this study is to characterize the safety, tolerability, pharmacokinetics (PK), Immunogenicity and preliminary antitumor activity of HC006 in subjects with advanced solid tumor malignancies. This study is a first-in-human (FIH) study of HC006 in subjects with advanced solid tumors.

DETAILED DESCRIPTION:
HC006, a novel therapeutic monoclonal antibody that specifically binds to human C-C motif chemokine receptor 8 (CCR8) and is designed to selectively deplete tumor-infiltrating T regulatory cells (Tregs) with enhanced antibody-dependent cell-mediated cytotoxicity (ADCC). In mouse tumor models, HC006 has demonstrated excellent antitumor activity and safety profile. This first-in-human (FIH) study will be conducted in two parts. In the Dose-Escalation part, testing will be done on up to 31 subjects to determine the maximum tolerated dose (MTD) and the recommended dose (RD). In the Dose-expansion part, we will evaluate the safety and efficacy of the recommended dose of HC006 in the treatment of advanced solid tumor subjects without standard therapy.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have histologically confirmed and documented diagnosis of locally advanced unresectable or metastatic advanced solid tumor that is refractory to standard treatment, or intolerant to standard treatment, or for which no standard treatment exists.
* At least one measurable disease for expansion cohorts per Response Evaluation Criteria in Solid Tumours (RECIST) v1.1(dose escalation only requires at least one assessable lesion)
* Agree to provide archived or fresh tumor tissue samples of primary or metastatic lesions for expansion cohorts.
* Life expectancy ≥12 weeks
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
* Have adequate organ function as described in the protocol.
* Agree to adopt effective contraceptive measures.

Exclusion Criteria:

* Prior exposure to CCR8 inhibitor or hypersensitivity to any ingredient of the study drug.
* Treatment with any systemic anti-cancer treatment within 4 weeks before first dose of study drug.
* Use of any live attenuated vaccines within 28 days.
* With primary central nervous system (CNS) tumors or unstable CNS metastases.
* Have active or history of autoimmune disease or immunodeficiency disease.
* With active, uncontrolled bacterial, viral, or fungal infections requiring systemic therapy.
* With any mental or cognitive impairment that may limit their understanding, implementation.
* Major surgery within 4 weeks of study drug administration.
* Have uncontrolled or severe illness, including but not limited to severe cardiovascular disease, interstitial lung disease or non-infectious pneumonia, or uncontrollable clinical third luminal effusion.
* Any adverse event from prior anti-tumor therapy has not yet recovered to ≤ grade 1 of CTCAE v5.0.
* History of other malignancy within the last 5 years, except for appropriately treated carcinoma in situ of the cervix, non-melanoma skin carcinoma.
* Women who are pregnant or breastfeeding.
* Other protocol defined exclusion criteria may apply.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Estimated)
Dates: Start 2024-02-27 (Actual); Primary Completion 2026-03-15 (Estimated); Study Completion 2026-07-16 (Estimated)

PRIMARY OUTCOMES:
Number of participants with Dose Limiting Toxicities(DLTs)as assessed by protocol | up to 24 months
  Incidence of Dose Limiting Toxicities(DLTs)
Number of participants with adverse events(AEs) as assessed by CTCAE v5.0 | up to 24 months
  Incidence of adverse events(AEs)
Number of participants with Serious adverse events(SAEs)as assessed by CTCAE v5.0 | up to 24 months
  Incidence of Serious adverse events(SAEs)
Percentage of Participants Experiencing Laboratory and ECG Abnormalities According to the NCI CTCAE v5.0 | up to 24 months
  Percentage of Participants Experiencing Laboratory and ECG Abnormalities According to the NCI CTCAE v5.0

SECONDARY OUTCOMES:
Pharmacokinetic (PK) Parameter:Maximum serum concentration (Cmax) | up to 24 months
  Maximum serum concentration (Cmax)
PK Parameter:Time to reach Cmax (Tmax) | up to 24 months
  Time to reach Cmax (Tmax)
PK Parameter:Area Under the Concentration-time Curve (AUC) | up to 24 months
  Area Under the Concentration-time Curve (AUC)
Immunogenicity | up to 24 months
  Incidence of anti-drug antibodies (ADAs) to HC006
Objective Response Rate (ORR) per RECIST 1.1 | up to 24 months
  The sum of the proportions of subjects who achieved CR or PR in imaging evaluation as assessed by the investigator based on RECIST1.1 criteria.
progression-Free Survival (PFS) per RECIST 1.1 | up to 24 months
  Time from first dose of the investigational drug to PD or death from any cause.
Overall Survival (OS) | up to 24 months
  Time from first dose of the investigational drug to death from any cause.
Disease Control Rate (DCR) per RECIST 1.1 | up to 24 months
  The sum of proportions of subjects who achieved CR, PR, and SD in imaging evaluation.
Duration of response (DOR) per RECIST 1.1 | up to 24 months
  Time from the first evaluated CR or PR until PD or death from any cause.
Time to progression (TTP) per RECIST 1.1 | up to 24 months
  Time from first dose of the investigational drug to the tumor evaluation of PD.
Time To Response (TTR) per RECIST 1.1 | up to 24 months
  Time from first dose of the investigational drug to the first tumor evaluation of CR or PR.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai East Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No